CLINICAL TRIAL: NCT02289261
Title: A Comparison of Morphine and Morphine Plus Dexmedetomidine in Chronic Cancer Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ersel GULEC, Ersel Gulec, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDICP01
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Morphine; Dexmedetomidine
MeSH Terms: conditions — Chronic Pain | interventions — Morphine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Morphine, 0.02 mg/kg PCA bolus dose with 10 minutes lock-out interval
  Interventions: Drug: Morphine
- Morphine plus dexmedetomidine (Active Comparator): Morphine 0.02 mg/kg plus dexmedetomidine 0.1 microgram/kg PCA bolus dose with 10 minutes lock-out interval
  Interventions: Drug: Morphine plus dexmedetomidine

INTERVENTIONS:
Drug: Morphine — Morphine, 0.02 mg/kg PCA bolus dose with 10 minutes lock-out interval
  Other Names: morphine sulphate
  Arms: Control
Drug: Morphine plus dexmedetomidine — Morphine 0.02 mg/kg plus dexmedetomidine 0.1 microgram/kg PCA bolus dose with 10 minutes lock-out interval
  Other Names: Morphine sulphate plus dexmedetomidine
  Arms: Morphine plus dexmedetomidine

SUMMARY:
The purpose of this study is to determine whether dexmedetomidine added to morphine is effective in the treatment of chronic cancer pain.

DETAILED DESCRIPTION:
We conduct the study in Cukurova University Faculty of Medicine Research Hospital after obtaining ethics committee approval and patient's informed consent. Patients with cancer pain are allocated into two group to receive Patient Controlled Analgesia with morphine or morphine plus dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic cancer pain
* between 20-80 years old age

Exclusion Criteria:

* the presence of severe systemic disease(cardiac, pulmonary, hepatic or renal)
* psychiatric or neurologic disease
* unable to communicate verbally
* nausea and vomiting
* patient's refusal

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Morphine consumption (mg) | 24 hours
  cumulative morphine consumption for 24 hours

SECONDARY OUTCOMES:
Pain score | 24 hours
  visual analog scale to assess pain degree

CONTACTS AND LOCATIONS:
Overall Officials: Selcuk Gök, M.D, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University Faculty of Medicine Research Hospital, Adana, Turkey (Türkiye)

REFERENCES:
- [Background] Blaudszun G, Lysakowski C, Elia N, Tramer MR. Effect of perioperative systemic alpha2 agonists on postoperative morphine consumption and pain intensity: systematic review and meta-analysis of randomized controlled trials. Anesthesiology. 2012 Jun;116(6):1312-22. doi: 10.1097/ALN.0b013e31825681cb. PMID 22546966
- [Result] Lin TF, Yeh YC, Lin FS, Wang YP, Lin CJ, Sun WZ, Fan SZ. Effect of combining dexmedetomidine and morphine for intravenous patient-controlled analgesia. Br J Anaesth. 2009 Jan;102(1):117-22. doi: 10.1093/bja/aen320. Epub 2008 Nov 5. PMID 18987053